CLINICAL TRIAL: NCT06216691
Title: Smart Phone Delivered Cognitive Behavioral Therapy for Adults With Psoriasis and Co-Morbid Depression Symptoms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Psoriasis Foundation (Other)
Responsible Party: Principal Investigator, John Barbieri, Assistant Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023P001944
Record Dates: First submitted 2024-01-12; First posted 2024-01-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis; Depressive Symptoms
MeSH Terms: conditions — Psoriasis; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Coach-guided smartphone delivered CBT program (Other): All eligible participants will be enrolled in an 8-week coach-guided smartphone delivered CBT program. The full duration of the program, with follow-up interview, will be 9 weeks.
  Interventions: Other: Coach-guided smartphone delivered CBT program.

INTERVENTIONS:
Other: Coach-guided smartphone delivered CBT program. — All eligible participants will be enrolled in an 8-week coach-guided smartphone delivered CBT program. The full duration of the program, with follow-up interview, will be 9 weeks.

SUMMARY:
A single arm, pilot study in which all eligible participants will be enrolled in an 8-week coach-guided smartphone delivered CBT program. The full duration of the program, with follow-up interview, will be 9 weeks.

DETAILED DESCRIPTION:
1. To demonstrate the feasibility and acceptability of coach-guided, smartphone-delivered CBT for depression among adults with psoriasis
2. To demonstrate the preliminary efficacy of coach-guided, smartphone-delivered CBT on the symptoms of depression and psoriasis

Primary endpoints

* Percentage of participants who engage with at least 6/8 (75%) modules
* Median Client Satisfaction Questionnaire-8 score at week 8
* Change from baseline in PHQ-9 at week 8

Secondary Endpoints

* Rate of participant dropout
* App acceptability to participants, as measured by the uMARS
* Change from baseline in Skindex-16 at week 8
* Change from baseline in PSI at week 8
* Change from baseline in AAI at week 8
* Frequency & severity of related adverse events
* The patient perspective on the feasibility and acceptability (qualitative)

Analysis Plan Investigators will assess the feasibility of smartphone-based CBT by reporting the proportion of participants who engaged with at least 75% of the treatment modules and assess patient acceptability with descriptive statistics summarizing the Client Satisfaction Questionnaire scores. Paired t-tests will be used to examine the differences in the pre- and post- treatment PHQ-9 scores, in all patients who complete the baseline study visit. Additionally, secondary outcomes (dropout rates, patient feedback from the Mobile Application Rating Scale, Skindex-16, Psoriasis Symptom Inventory, Appearance Anxiety Inventory) will be reported descriptively. Post-treatment interviews will be transcribed, edited for clarity, coded to identify themes and summarized.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 18 years of age and older

  * Dermatologist confirmed diagnosis of psoriasis
  * Current depression symptoms, defined as a PHQ-9 score of 5 or greater
  * Current psoriasis symptoms, defined as a scaled score of "mild" on any of the Skindex-16 subscales
  * Participants must be proficient in English and have access to an Android or iOS smartphone

Exclusion Criteria:

* Previous participation in CBT for depression
* Current participation in any type of psychotherapy
* Those on psychotropic medications must be taking a stable dose for 2 months prior to enrollment and be willing to remain at a stable dose during the 8-week study
* Current elevated suicide risk (see Section 5.3 for details)
* Individuals who are incarcerated or compulsory detained
* Any uncontrolled or poorly controlled chronic medical condition that may interfere with an individual's ability to participate in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants Engagement | from Baseline to 8 Weeks
  Percentage of participants who engage with at least 6/8 (75%) modules within the app
Client Satisfaction Questionnaire-8 (CSQ-8) | change from baseline to Week 8
  The CSQ-8 is an 8 item, self-reported questionnaire that measures satisfaction with clinical services received on a 1-4 scale. Scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction .
Patient Health Questionaire-9 (PHQ-9) | Week 8
  The PHQ-9 is a widely used, reliable, and valid self-report measure of depression severity, It includes nine Likert scale items ranging from 0 (not at all) to 3 (every day), where higher scores indicate more severe depressive symptoms.

SECONDARY OUTCOMES:
Rate of participant dropout | Week 8
  Amount of participants do not complete the study
user Mobile Health Rating Scale (uMARS) | Week 8
  The uMARS is a 20-item measure provides reliable measure of app quality in target users. It includes 4 objective quality subscales-engagement, functionality, aesthetics, and information quality and 1 subjective quality subscale. Each feature is rated on a scale from 1 (inadequate) to 5 (excellent).
Skindex-16 | Week 8
  The Skindex-16 is a brief patient reported outcome that measures functioning, emotions and symptoms associated with chronic skin diseases. Each item is assessed on a 7-point Likert scale and all responses are transformed to a linear scale of 100. The over all score ranges from 0 (no effect) to 100 (effect experienced all the time).
Appearance Anxiety Inventory (AAI) | Week 8
  The AAI is a 10 item self-report questionnaire assessing the frequency of cognitive processes (e.g., rumination, self-focused attention) and behavioral responses (e.g. social avoidance, appearance checking) in Body Dysmorphic Disorder (BDD). Individuals respond to items on a 5-point Likert Scale (0= not all to 4= all the time) and a total score is obtained by summing all the items (range is 0 to 40). The reliable change score is 7 and above.
Frequency of participants with adverse events | Week 8
  Participants will be asked to describe any new health problems or injuries and developed while participanting in the study.
Psoriasis Symptom Inventory | Week 8
  ): The PSI is an eight-item patient-reported outcome measure for assessing severity of plaque psoriasis symptoms including itch, redness, scaling, burning, cracking, stinging, flaking, and pain). Each item is scored on a 5-point Likert scale where high score indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States